CLINICAL TRIAL: NCT04949542
Title: Development and Testing of a Caregiver-facing Mobile Health Intervention to Reduce Duration of Untreated Psychosis
Brief Title: Bolster: Caregiver App to Reduce Duration of Untreated Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Benjamin Buck, Assistant Professor: School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00013334
Record Dates: First submitted 2021-06-17; First posted 2021-07-02 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Caregiver to a Young Adult With Early Psychosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolster (Experimental): Participants in the experimental arm will be provided access to the Bolster smartphone application designed to support caregivers of young adults with early psychosis as well as the support resources offered in the control condition. They will also have access to the research team by phone for technical troubleshooting and support as necessary.
  Interventions: Behavioral: Bolster
- Control (Other): Participants in the control condition will be provided support resources from mental health advocacy organizations representing currently available resources for caregivers (including a selection from the National Alliance on Mental Illness and Mental Health America). They will also have access to the research team by phone for technical troubleshooting and support as necessary.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Bolster — Bolster is a native mobile app that provides on-demand content to caregivers of young adults with early psychosis to support their caregiving skills and knowledge of psychosis.
  Arms: Bolster
Behavioral: Control — Exemplar resources provided in the control arm will include a selection from the National Alliance on Mental Illness and Mental Health America designed to support caregivers helping loved ones access care.
  Arms: Control

SUMMARY:
The proposed research project aims to develop and test a mobile health intervention designed to improve caregivers' illness knowledge and caregiving skills through interactive cognitive-behavioral modules, and through these improvements, reduce distress, improve coping, improve family communication, increase caregiver treatment facilitation and reduce duration of untreated psychosis. This clinical trial will involve a remote pilot randomized controlled trial comparing this new intervention to existing online caregiving support resources. Analyses will determine whether this approach is acceptable and feasible, as well as explore its effectiveness and impact on key components of the cognitive model of caregiving.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Live in the United States
* Caregiver to a young adult with early psychosis, wherein early psychosis is defined as: (1) Being between the ages of 15 and 35, and (2) Within the past five years, the young adult first experienced: (2A) Presence of psychotic symptoms represented by one or more of hallucinations, delusions, marked thought disorder, psychomotor disorder or bizarre behavior, as well as (2B) Definite change of personality or behavior manifesting as two or more of the following: serious deterioration of function, marked social withdrawal, persistent self-neglect, episodic marked anxiety.
* A positive screen according to the Caregiver Prime Screen - Revised (endorsed two or more responses of five or six ("somewhat"/"definitely" agree))
* Own an Apple iPhone
* Self-identify as a caregiver of the affected person
* The affected person is not enrolled in specialty mental health services (i.e. a program wherein the affected person can access psychiatry and counseling/therapy services), and has not been enrolled in such services for at least three months prior to screening. If an affected person is receiving one of these services, the caregiver reports that this is an inadequate level of care.

Exclusion Criteria:

* Incarceration or long-term care setting for either the caregiver or identified affected young adult.
* Participant failed to demonstrate understanding of study details in comprehension screening process.
* The affected person is unengaged in services, but only as a result of having completed or "graduated" from a specialty treatment program for psychosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Buck, PhD, Principal Investigator — University of Washington
Locations (1):
- Behavioral Research in Technology and Engineering Center, Health Sciences, UW Medical Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bolster | Control
Started | 40 | 20
Completed | 36 | 19 (One participant did not complete the post-test assessment, but provided partial data, therefore for some outcome measures, this number is N = 20 at post-test.)
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bolster | Control | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.73 (7.26) | 54.40 (8.31) | 54.62 (7.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 19 | 56
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 37 | 18 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Black or African American | 4 | 1 | 5
  More than one race | 1 | 0 | 1
  Other | 2 | 0 | 2
  White | 30 | 18 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Family Communication
Description: Family communication will be assessed with the Family Questionnaire (FQ). The FQ is a 20-item self-report assessment of criticism and emotional expression in interactions with family members toward patients with mental illness. Each item is rated on a 4-point scale (1 = never/very rarely; 4 = very often). The FQ is scored by summing individual items with higher scores indicating greater levels of expressed emotion. As a primary outcome, we will examine the combined total of emotional overinvolvement and critical comments; scores range from 20 to 80 with higher scores indicating greater expressed emotion.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 58.94 (8.36) | 56.66 (6.82)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 53.23 (8.74) | 53.20 (9.09)
  12 weeks: number analyzed (Participants) | 36 | 20
  12 weeks | 52.02 (8.43) | 53.55 (8.31)

2. Primary Outcome: Change in Treatment Facilitation
Description: Treatment seeking will be measured using the Measure to Assess Steps to Service-Caregivers (MASS-CG). The MASS-CG is a 23-item self-report assessment of steps taken by the caregiver towards the attainment of mental health treatment for their loved one, including research, social support, encouragement or support of the loved one's help-seeking actions, and engagement with service provider steps. Each item is endorsed on a three-point Likert scale (0 = No, I have not done this, 1 = I have done this once or twice, 2 = I have done this multiple times). The MASS-CG is scored by summing individual items with higher scores indicating greater levels of treatment facilitation activities.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline: number analyzed (Participants) | 40 | 19
  Baseline | 22.47 (9.97) | 24.29 (13.89)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 18.79 (10.08) | 16.60 (8.86)
  12 weeks: number analyzed (Participants) | 36 | 20
  12 weeks | 20.08 (9.62) | 19.54 (11.16)

3. Primary Outcome: Change in Loved One Treatment Engagement, Medication Provider
Description: Treatment facilitation / duration of untreated psychosis will be assessed according to participants' report of appointments attended by their relative in the past during the treatment period. This first category includes meeting with a clinician providing psychiatric medications. At screening, participants report treatment engagement over the previous three months and during the study period, participants are asked to report on this weekly. This count variable represents the number of participants who reported that their loved one attended an appointment with a medication provider in the three months preceding the study period reported at screening ("Baseline") as well as for the duration of the study period reported in weekly brief assessments ("12 weeks"). The 12 week data point includes participants who completed at least half of the weekly brief assessments.
Time Frame: Baseline, 12 weeks
Population: Participants are included in the 12 week total if they completed more than half the brief assessments during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
Participants
  Baseline | 15 | 8
  12 weeks: number analyzed (Participants) | 38 | 20
  12 weeks | 21 | 7

4. Primary Outcome: Change in Loved One Treatment Engagement, Therapy or Counseling
Description: Treatment facilitation / duration of untreated psychosis will be assessed according to participants' report of appointments attended by their relative in the past during the treatment period. This first category includes meeting with a clinician providing mental health therapy or counseling. At screening, participants report treatment engagement over the previous three months and during the study period, participants are asked to report on this weekly. This count variable represents the number of participants who reported that their loved one attended an appointment for psychotherapy or counseling in the three months preceding the study period reported at screening ("Baseline") as well as for the duration of the study period reported in weekly brief assessments ("12 weeks"). The 12 week data point includes participants who completed at least half of the weekly brief assessments.
Time Frame: Baseline, 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
Participants
  Baseline | 17 | 8
  12 weeks: number analyzed (Participants) | 38 | 20
  12 weeks | 24 | 8

5. Secondary Outcome: Change in Illness Knowledge, Factual Knowledge
Description: This is assessed with the Knowledge About Schizophrenia (KAST), an 18-item multiple-choice assessment examining individuals' knowledge of the etiology, symptoms, and prognosis of schizophrenia. Total scores indicate the number of correct responses, and thus range from 0 to 18.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 15.90 (2.25) | 15.65 (1.53)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 16.16 (1.54) | 16.15 (1.53)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 16.08 (1.79) | 15.63 (1.95)

6. Secondary Outcome: Change in Illness Knowledge, Caregiver Self-rated
Description: Illness appraisals will be assessed with the Illness Perception Questionnaire for Schizophrenia Relatives (IPQSR), a self-report scale of caregivers' beliefs about the severity, prognosis, and responsiveness to treatment of mental illnesses. Each item is rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree), and totals are scored by summing individual items. For the coherence total, we are totaling the 5 items related to the caregiver's report of how much they understand or know about their loved one's illness. Scores range from 5 to 25 with lower scores indicating better self-rated understanding or coherence.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 13.40 (3.56) | 11.35 (4.18)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 10.97 (3.27) | 10.96 (4.21)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 10.92 (3.21) | 10.58 (3.40)

7. Secondary Outcome: Change in Illness Appraisals, Consequences
Description: Illness appraisals will be assessed with the Illness Perception Questionnaire for Schizophrenia Relatives (IPQSR), a self-report scale of caregivers' beliefs about the severity, prognosis, and responsiveness to treatment of mental illnesses. Each item is rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree), and totals are scored by summing individual items. For the consequences total, we are totaling the 20 items related to consequences affecting the caregiver and the affected person. Scores range from 20 to 100 with higher scores indicating greater perceptions of negative consequences.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 79.63 (9.60) | 80.90 (12.46)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 76.13 (9.89) | 79.77 (12.71)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 75.93 (11.93) | 80.39 (10.70)

8. Secondary Outcome: Change in Illness Appraisals, Control
Description: Illness appraisals will be assessed with the Illness Perception Questionnaire for Schizophrenia Relatives (IPQSR), a self-report scale of caregivers' beliefs about the severity, prognosis, and responsiveness to treatment of mental illnesses. Each item is rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree), and totals are scored by summing individual items. For the control total, we are totaling the 8 items related to caregiver, affected person, and treatment control over illness course. Scores range from 8 to 40 with higher scores indicating greater perceptions of possibilities for actions that affect the course of illness.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
units on a scale
  Baseline | 30.06 (4.18) | 31.70 (4.23)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 30.65 (4.73) | 31.80 (4.07)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 31.46 (4.46) | 31.63 (4.03)

9. Secondary Outcome: Change in Illness Appraisals, Emotional Distress About Illness
Description: Illness appraisals will be assessed with the Illness Perception Questionnaire for Schizophrenia Relatives (IPQSR), a self-report scale of caregivers' beliefs about the severity, prognosis, and responsiveness to treatment of mental illnesses. Each item is rated on a 5-point scale (1 = strongly disagree; 5 = strongly agree), and totals are scored by summing individual items. For the emotional distress score, we are examining the emotional representation scale, a 9-item scale with scores ranging from 9 to 45, with higher scores indicating greater emotional distress.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 34.74 (6.39) | 31.85 (6.28)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 30.63 (5.30) | 32.55 (5.63)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 29.64 (6.47) | 32.11 (8.15)

10. Secondary Outcome: Change in Appraisal of Caregiving Experiences**
Description: Appraisals of caregiving experiences will be assessed with the Brief Experience of Caregiving Inventory (BECI).** The BECI is a 19-item assessment of the impact of caregiving on the individual's life, both in negative and positive ways. The items are rated on a 5-point Likert scale (never to nearly always), and scores range from 0 to 76, with a higher score denoting more negative appraisals of one's caregiving experience.
  **NOTE: The version of the BECI that was administered used instructions asking participants to report on their experiences in the month following their loved one's first hospitalization. Due to this, this measure is best interpreted as caregivers' changing appraisals of their early experiences of caregiving. There was also heterogeneity in participants' report of their loved one ever having experienced a hospitalization in our sample that also affects interpretation of this measure.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline: number analyzed (Participants) | 39 | 20
  Baseline | 43.04 (11.08) | 45.77 (11.24)
  6 weeks: number analyzed (Participants) | 36 | 20
  6 weeks | 40.11 (11.91) | 42.70 (14.46)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 37.94 (10.92) | 42.76 (12.26)

11. Secondary Outcome: Change in Caregiver Coping, Activities
Description: Caregiver coping will be assessed with the Brief COPE Inventory, a 28-item self-report scale of coping skills in response to stressors, based on the full COPE inventory; items generate a range of subscale scores related to specific coping areas. The instrument consists of 28 items which will be scored on a 1 to 4 Likert scale (I haven't been doing this at all to I've been doing this a lot), with higher values representing a greater frequency of engaging in each coping strategy. For this outcome, we will examine total frequency sum of items (14) assessing variables a priori selected to represent adaptive coping. Scores on this scale range from 14 to 56.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 35.32 (6.06) | 37.25 (6.21)
  6 weeks: number analyzed (Participants) | 36 | 20
  6 weeks | 36.07 (7.30) | 34.72 (7.30)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 36.81 (7.80) | 36.84 (6.58)

12. Secondary Outcome: Change in Caregiver Coping, Self-efficacy
Description: Caregiver coping self-efficacy will be assessed with the Coping Self-Efficacy Scale, a 26-item self-report questionnaire measuring the perceived ability of coping with various life challenges. Responses are rated on a 0 to 10 scale, and scores range from 0 to 260, with higher scores denoting a greater sense of self-efficacy in coping.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 135.23 (42.06) | 142.23 (40.85)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 154.86 (38.90) | 149.25 (44.57)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 168.99 (42.22) | 160.84 (44.89)

13. Secondary Outcome: Change in Caregiver Distress
Description: Caregiver distress (secondary mediator) will be assessed with General Health Questionnaire (GHQ), a 12-item questionnaire assessing general psychological morbidity. Respondents indicate agreement on a four-point scale (0 = Not at all; 3 = More than usual) and total scores ranging from 0 to 36 with higher scores indicating more severe psychological morbidity.
Time Frame: Baseline, 6 weeks, 12 weeks
Population: Participants are only analyzed (and total scores mean imputed) if they completed more than half the items on the scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bolster | Control
Number analyzed (Participants) | 40 | 20
score on a scale
  Baseline | 19.00 (6.48) | 18.45 (8.68)
  6 weeks: number analyzed (Participants) | 37 | 20
  6 weeks | 14.14 (6.18) | 17.75 (9.03)
  12 weeks: number analyzed (Participants) | 36 | 19
  12 weeks | 11.67 (6.43) | 15.68 (8.85)

ADVERSE EVENTS:
Time Frame: Full duration of study period, 12 weeks
Arm/Group | Bolster | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT04949542/Prot_SAP_000.pdf